CLINICAL TRIAL: NCT03034382
Title: Adjuvants to Ultrasonic Guided Interscalene Block In Arthroscopic Rotator Cuff Repair; Morphine and/or Nalbuphine
Brief Title: Morphine and/or Nalbuphine as Adjuvants in Ultrasound Guided Interscalene Block: for Shoulder Surgeries
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Abbas Hassan, Primary investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SH1
Record Dates: First submitted 2017-01-19; First posted 2017-01-27 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Rotator Cuff Tear
Keywords: morphine; nalbuphine; arthroscopic rotator cuff repair; ultrasound guided interscalene block
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Morphine; Nalbuphine; Bupivacaine; Lidocaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (4):
- Morphine (Experimental): 5 mg morphine in 5ml volume injected as adjuvants to 10 ml of lidocaine and epinephrine 1:400,000.
  Interventions: Drug: Morphine; Drug: Lidocaine Hydrochloride 1% and epinephrine 1:400,000
- Nalbuphine (Experimental): 5 mg nalbuphine in 5ml volume injected as adjuvants to 10 ml of lidocaine and epinephrine 1:400,000.
  Interventions: Drug: Nalbuphine; Drug: Lidocaine Hydrochloride 1% and epinephrine 1:400,000
- Morphine and Nalbuphine (Experimental): 5 mg morphine and 5 mg nalbuphine in 5 ml volume are injected as adjuvants to 10 ml of lidocaine and epinephrine 1:400,000.
  combination of 5 mg morphine and 5 mg nalbuphine in 5 ml volume are injected perineurally as adjuvants for 10 ml of lidocaine + epinephrine 1:400,000 in ultrasound guided interscalene block
  Interventions: Drug: Morphine; Drug: Nalbuphine; Drug: Lidocaine Hydrochloride 1% and epinephrine 1:400,000
- Bupivacaine 0.5% (Placebo Comparator): 10 ml of lidocaine 1% and epinephrine 1:400,000 and 5 ml of Bupivacaine 0.5% in interscalene block.
  Interventions: Drug: Bupivacaine 0.5%; Drug: Lidocaine Hydrochloride 1% and epinephrine 1:400,000

INTERVENTIONS:
Drug: Morphine — 5 mg morphine in 5 ml volume are injected perineurally as adjuvants for 10 ml of lidocaine + epinephrine 1:400,000 in ultrasound guided interscalene block
  Other Names: morphine sulphate
  Arms: Morphine; Morphine and Nalbuphine
Drug: Nalbuphine — 5 mg nalbuphine in 5 ml volume are injected perineurally as adjuvants for 10 ml of lidocaine + epinephrine 1:400,000 in ultrasound guided interscalene block
  Other Names: nubain
  Arms: Morphine and Nalbuphine; Nalbuphine
Drug: Bupivacaine 0.5% — 10 ml of 1% lidocaine +1:400,000 epinephrine and 5 ml of bupivacaine 0.5% injected perineurally in interscalene block
  Other Names: Marcaine HCL
  Arms: Bupivacaine 0.5%
Drug: Lidocaine Hydrochloride 1% and epinephrine 1:400,000 — 10 ml of 1% lidocaine and 1:400,000 epinephrine were injected perineurally in interscalene block
  Other Names: lidocaine HCL and Adrenaline

SUMMARY:
the aim of this study is to evaluate the duration of analgesia when either morphine or nalbuphine or both are used as adjuvants in sonar guided interscalene brachial plexus block for arthroscopic rotator cuff repair.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for arthroscopic repair of rotator cuff muscle tear of the shoulder.
* ASA physical status I - Ш.

Exclusion Criteria:

* Infection at the site of injection.
* Coagulopathy or other bleeding diathesis.
* Known allergy to drugs in the study
* Preexisting neurologic deficits in the area to be blocked.
* Inability to communicate with the investigator and the hospital staff.
* History of chronic opioid use.
* Morbid obesity BMI>40.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
the total number of analgesic requests | 72 hours postoperative followup
  the combination of opioid agonist and mixed agonist-antagonist peripherally prevents the development of early tolerance of the opioid agonist; thus the agonist would maintain the same efficacy and this will be obvious clinically by a reduction in the requests for supplementary analgesia.

SECONDARY OUTCOMES:
duration of analgesia | 72 hours followup
  duration of analgesia when morphine or nalbuphine or both used in interscalene block using VAS.
patient satisfaction | 72 hours followup
  - The patient satisfaction score. Patients were also asked to rate their satisfaction with the analgesia on a scale of 0-10 (0 for total dissatisfaction to 10 for total satisfaction).
The first time to ask for analgesics | 72 hours followup
sedation score | 72 hours followup
  recorded every 4 hours; ranging from alert, drowsy, sleeping but responsive to verbal commands up to unarousable (we consider sedation score 3 or more as clinically significant sedation that mandate close patient observation every hour).
number of vomiting attacks | 72 hours followup
  recorded every 4 hours. A vomiting attack was defined by events of vomiting that occurred in a rapid sequence (<1 minute between events). If vomiting was separated by more than 1 minute; they will be considered to be separate attacks. Retching (the same as vomiting but without expulsion of gastric contents) was considered as vomiting. If the patient experienced vomiting; ondansetron 4 mg IV was given.
itching | 72 hours followup
  Itching is assessed using an ordinal scale (0 = no itch, 1 = mild, 2 = moderate, 3 = severe).

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud A Aly, Prof, Study Chair — Assiut University Hospitals; Kawser H Mohammed, Prof, Study Chair — Assiut University Hospitals; Ayman A Mamdouh, Ass Prof, Study Director — Assiut University Hospitals
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided